CLINICAL TRIAL: NCT00114933
Title: Phase III-IV, Comparative, Randomized, Open-Label, Study to Evaluate Safety and Efficacy of Suspending Nucleosides From a Triple-Drug Therapy Based on Lopinavir/Ritonavir Versus Continuing Triple-Drug Therapy in HIV-Infected Subjects With Undetectable Plasma HIV Viremia for Six Months
Brief Title: "OK 2004 Study" (Only Kaletra 2004 Study): Study to Evaluate Suspending Nucleosides From Triple-Drug Therapy in HIV Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arribas, Jose R., M.D. (Individual)
Collaborators: Pulido, Federico, M.D. (Individual); Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPA-378-05-40; EudraCT 2004-001323-37
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: Stopping nucleosides and continuing lopinavir/ritonavir monotherapy

SUMMARY:
Lopinavir/ritonavir monotherapy may maintain virologic suppression in patients who have been undetectable for six months while on triple drug antiretroviral therapy. Lopinavir/ritonavir pharmacokinetics might prevent resistance development in patients who experience virological rebound after single-drug simplification.

DETAILED DESCRIPTION:
Primary Study Objective: Efficacy and durability of switching to lopinavir/ritonavir single-drug HAART compared to maintaining therapy based on lopinavir/ritonavir and two nucleosides

Secondary Study Objective(s):

* Safety (related drug AEs/SAEs and laboratory anomalies G3/4) through 48 w.
* Resistance profile on patients with sustained virological failure
* QOL comparing stopping nucleosides versus continuing therapy
* Pharmaco-economic analysis comparing treatment cost between the 2 study arms.
* Predicting factors of failure in the stopping nucleosides arm

Subject Population: 200 patients

Study Design:

RANDOMIZATION:

Patients are randomized (1:1) either to continue under the same treatment or stop nucleosides as follows:

* Stopping nucleosides arm: Lopinavir/r alone.
* Continuing arm: Lopinavir/r + 2 NRTIs

STUDY PROCEDURES: A baseline HIV-RNA, CD4 and routine labs will be collected if the most recent results are not collected within the 4 weeks prior entering the study. Patients will be followed for HIV-RNA (and CD4) at w1, w4, w8, w16, w24, w 36 and w48. After w48, durability of response to lopinavir/r single-drug therapy will be studied long-term (up to w96). Routine hematology and clinical chemistry (including fasting triglycerides and cholesterol, total and HDL/LDL ratio) will be measured at w4, w16, w24, w 36 and w48. A central laboratory will be used for HIV-RNA determinations and to archive plasma/cell samples for further genotype test in case of rebound.

Treatment adherence will be followed with a self-patient report questionnaire (GEEMA study)

All AEs will be collected if suspected relation (possible or probable) to any concomitant ARV drug, and SAEs, related or not, reported within 24h.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients > 18 years old who provide signed and dated Informed consent.
* HIV patients who have been receiving lopinavir/ritonavir and two nucleosides during at least 4 weeks.
* Plasma HIV RNA < 50 cop/ml for six months

Exclusion Criteria:

* HIV patients who have stopped a protease inhibitor due to virological failure.
* HIV patients with hepatic or renal insufficiency.
* HIV patients with positive serum HBVAg
* HIV patients who require treatment with a lopinavir/r contraindicated medication.
* HIV pregnant or breastfeeding women.
* Active drug abuse (including alcohol or recreational drugs). Exception, cannabis, provided the investigator is confident in patient adherence. Patients under Methadone program will be accepted too if deemed appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2007-05

PRIMARY OUTCOMES:
% patients with therapeutic failure in both arms at 48 weeks (OT and ITT)

SECONDARY OUTCOMES:
% patients with virological failure: HIV-RNA > 500 cop/ml under the randomly assigned therapy (OT and ITT)
% patients with HIV RNA < 500 cop/ml and < 50 cop/ml at w24, w48 (OT and ITT)
Time to virological failure per Kaplan Meyer analysis
CD4 cell count change from baseline
Percentage of viruses with resistance in the protease gene at w24 and w48
Description of AEs with probable, possible or unknown relationship to study drug

CONTACTS AND LOCATIONS:
Overall Officials: José R. Arribas, MD, Study Chair — Hospital La Paz; Federico Pulido, MD, Study Chair — Hospital 12 de Octubre
Locations (28):
- Spain (28):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital General de Elche, Elche, Alicante
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Sant Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Insular, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital de Donostia, San Sebastián, Guipuzcoa
  - Hospital U. Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Xeral Cies, Vigo, Pontevedra
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Nuestra Señora de Valme (Sevilla), Seville, Sevilla
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Dr. Peset, Valencia, Valencia
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Arribas JR, Delgado R, Arranz A, Munoz R, Portilla J, Pasquau J, Perez-Elias MJ, Iribarren JA, Rubio R, Ocampo A, Sanchez-Conde M, Knobel H, Arazo P, Sanz J, Lopez-Aldeguer J, Montes ML, Pulido F; OK04 Study Group. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and 2 nucleosides for maintenance therapy of HIV: 96-week analysis. J Acquir Immune Defic Syndr. 2009 Jun 1;51(2):147-52. doi: 10.1097/QAI.0b013e3181a56de5. PMID 19349870
- [Derived] Pulido F, Arribas JR, Delgado R, Cabrero E, Gonzalez-Garcia J, Perez-Elias MJ, Arranz A, Portilla J, Pasquau J, Iribarren JA, Rubio R, Norton M; OK04 Study Group. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and two nucleosides for maintenance therapy of HIV. AIDS. 2008 Jan 11;22(2):F1-9. doi: 10.1097/QAD.0b013e3282f4243b. PMID 18097218